CLINICAL TRIAL: NCT02650154
Title: The Effects of the Anesthetic Ketamine in Young Children Undergoing Procedural Sedation
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Yaron Finkelstein, Staff Physician, The Hospital for Sick Children
Other Study IDs: REB1000033567
Record Dates: First submitted 2016-01-05; First posted 2016-01-08 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Trauma
Keywords: sedation; children; infants; ketamine; neurotoxicity
MeSH Terms: conditions — Wounds and Injuries; Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-ketamine group: Blood samples are taken prior to the administration of ketamine.
- Post-ketamine group: Blood samples are taken several hours after the administration of ketamine.

SUMMARY:
In the emergency department (ED), ketamine is a popular anesthetic agent during sedation of children for painful and other short procedures. Sedation for procedures is more commonly used in children than adults, to achieve motion control and cooperation. In children, ketamine offers an ideal choice due to the fact that it is short acting, a highly effective sedative, and preserves cardio-respiratory stability. In the United States, more than one million children per year up to four years of age undergo short procedures requiring anesthestic agents, including ketamine. However, there is mounting concern from animal studies and retrospective human research regarding the safety of ketamine when administered to infants and young children with respect to its potential toxic effects on the developing . Conversely, ketamine has also been suggested as a neuroprotective agent. Prompt investigation and resolution of this issue is urgently required.

DETAILED DESCRIPTION:
The objectives of this study are:

Primary Objective: In otherwise healthy children between 3 and 48 months of age who present to a tertiary care emergency department and receive procedural sedation with ketamine, to determine if there is at least a 50% increase, compared to baseline in the serum concentration of any of the neurotoxicity biomarkers S100B, glial fibrillary acidic protein (GFAP) or neuronal-specific enolase (NSE), 1 to 3 hours after intravenous ketamine administration. The cut-off of 50% is a benchmark value routinely quoted in both animal and human studies, which correlated neurotoxicity biomarker levels with functional outcomes.

Secondary Objectives: In the aforementioned population:

1. To determine if at least a 50% increase in the serum concentration of S100B, GFAP or NSE compared to baseline at 6 to 12 hours after intravenous ketamine administration.
2. To explore if genotypes relevant to ketamine metabolism and disposition are associated with increased vulnerability to the neurotoxic effects of ketamine.
3. To determine the toxic effect of ketamine administration at the cellular level (evidence of sustainable cellular damage and mitochondrial DNA changes).

ELIGIBILITY:
Inclusion Criteria:

1. All children between the ages of 3 and 48 months who receive intravenous ketamine for procedural sedation in the ED during study enrolment hours will be eligible for recruitment.

Exclusion Criteria:

1. Children with contraindications to procedural sedation in the ED according to SickKids (the Hospital for Sick Children) practice guidelines or to ketamine administration will not be considered.
2. Parents with an insurmountable language barrier (i.e. does not speak English and are not accompanied by another adult who cannot translate for the parent/caregiver), which prevents informed consent.
3. Child who has received procedural sedation/ or surgery under general anesthesia in the past 30 days.
4. A child who has received any central nervous system drugs (e.g. anticonvulsants, benzodiazepines) or a known neurotoxic drug (e.g., methotrexate, corticosteroids) concomitantly or in the 30 days preceding the sedation.
5. A child who has suffered traumatic head injury concomitantly or in the previous 30 days
6. A child who has CNS (Central Nervous System) illnesses or pathologies (e.g., meningitis, near drowning, hypoxic-ischemic brain injury, seizure disorder) in the 30 days prior to sedation, potentially leading to elevated baseline serum biomarkers.
7. A child whose parents are considered to be in emotional distress due to the injury or illness of the child by the attending ED physician or where the attending ED physician does not believe it is appropriate to ask the parents for consent.

Ages: 3 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children between the ages of 3 and 48 months who receive intravenous ketamine for procedural sedation in the ED during study enrolment hours will be eligible for recruitment.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Increase in serum biomarkers of neurotoxicity (neuronal cell apoptosis) | 1 to 24 hours from ketamine exposure

SECONDARY OUTCOMES:
Ketamine-induced mitochondrial damage | 1-24 hours from ketamine exposure
  Peripheral blood cells we be tested for for mitochondrial damage (changes in biomass and mtDNA) post ketamine exposure. Isolated lymphocytes from pre- and post-ketamine exposure blood samples from each patient will be split into two pools analysed for changes to mitochondrial content and mtDNA damage. The first pool will be stained with mitochondrial membrane potential-specific dye (TMRM) and imaged to reveal changes in mitochondrial morphology and function. DNA will be isolated from the second pool and probed for both cellular mitochondrial content and mtDNA damage using quantitative PCR (Polymerase Chain Reaction).
Pharmacogenetics role in ketamine toxicity | 1-24 hours from ketamine exposure
  In each patient we will determine the allele distribution (proportions/percentages) of polymorphic genes associated with the metabolism of ketamine.

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Finkelstein, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No